CLINICAL TRIAL: NCT03131453
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of CNP520 in Participants at Risk for the Onset of Clinical Symptoms of Alzheimer's Disease (AD).
Brief Title: A Study of CNP520 Versus Placebo in Participants at Risk for the Onset of Clinical Symptoms of Alzheimer's Disease
Acronym: GS2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to safety issues.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Amgen (Industry); Banner Alzheimer's Institute (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCNP520A2202J; 2016-002976-28 (EudraCT Number)
Record Dates: First submitted 2017-04-05; First posted 2017-04-27 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Alzheimers Disease
Keywords: Placebo controlled; APOE4 carriers; Homozygotes; Heterozygotes; Brain Amyloid; Aβ lowering; BACE-1 inhibitor; CNP520; elderly; preclinical Alzheimers disease; Alzheimers Disease; Prevention; Unimpaired cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — Umibecestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CNP520 50 mg (Experimental): 50 mg capsule taken orally once daily
  Interventions: Drug: CNP520 50mg
- CNP520 15 mg (Experimental): 15 mg capsule taken orally once daily
  Interventions: Drug: CNP520 15mg
- Placebo (Placebo Comparator): Matching placebo to 15 and 50 mg CNP520 taken orally once daily
  Interventions: Other: Matching placebo

INTERVENTIONS:
Drug: CNP520 50mg — 50 mg capsule
  Arms: CNP520 50 mg
Drug: CNP520 15mg — 15 mg capsule
  Arms: CNP520 15 mg
Other: Matching placebo — Matching placebo for 15 and 50 mg capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of CNP520 on cognition, global clinical status, and underlying AD pathology, as well as the safety of CNP520, in people at risk for the onset of clinical symptoms of AD based on their age, APOE genotype and elevated amyloid.

DETAILED DESCRIPTION:
This trial was a randomized, double-blind, placebo-controlled, parallel group, adaptive design with variable treatment duration planned in cognitively unimpaired participants aged 60 to 75 years, with at least one apolipoprotein E allele (APOE4), (homozygotes (HMs) or heterozygotes (HTs)) and, if HTs, with evidence of elevated brain amyloid. The participants were randomized to either CNP520 50 mg, CNP520 15 mg or placebo a 2:1:2 ratio and was stratified based on amyloid status. The planned treatment period of 5 to 8 years was not achieved due to early study termination.

ELIGIBILITY:
Inclusion Criteria:

* consent to receive disclosure of their risk estimates to develop clinical symptoms of AD based on their APOE genotype and, if Heterozygotes, evidence of elevated brain amyloid.
* Male or female, age 60 to 75 years inclusive. Females must be considered post-menopausal and not of child bearing potential
* Cognitively unimpaired as evaluated by memory tests performed at screening.
* Participant's willingness to have a study partner.
* Carrier of at least one APOE4 gene if Heterozygotes, elevated brain amyloid (as measured by CSF Abeta or amyloid PET imaging).

Exclusion Criteria:

* Any disability that could have prevented the participants from completing all study requirements. -
* Current medical or neurological condition that could have impacted cognition or performance on cognitive assessments.
* Advanced, severe progressive or unstable disease that could have interfered with the safety, tolerability and study assessments, or put the participant at special risk.
* History of malignancy of any organ system, treated or untreated, within the past 60 months.
* Indication for, or current treatment with ChEIs and/or another AD treatment (e.g. memantine).
* Contraindication or intolerance to MRI.
* Brain MRI results showing findings unrelated to AD that, in the opinion of the Investigator might be a leading cause to future cognitive decline, could have posed a risk to the participant, or could have prevented a satisfactory MRI assessment for safety monitoring.
* Suicidal Ideation in the past six months, or Suicidal Behavior in the past two years.
* A positive drug screen at Screening, if, in the Investigator's opinion, was is due to drug abuse.
* Significantly abnormal laboratory results at Screening, not as a result of a temporary condition.
* Current clinically significant ECG findings.
* Clinically relevant depigmenting or hypopigmenting conditions (e.g. albinism, vitiligo) or active / history of chronic urticaria in the past year.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (182):
- United States (90):
  - Banner Alzheimer's Institute, 901 East Willetta Street, Phoenix, Arizona
  - Banner Sun Health Research Institute, 10515 West Santa Fe Drive, Building B, Sun City, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - ATP Clinical Research Inc, 3151 Airway Avenue T 3, Costa Mesa, California
  - Irvine Center for Clinical Res, 2515 McCabe Way, Irvine, California
  - Torrance Clinical Research Institute, 25043 Narbonne Avenue, Lomita, California
  - Novartis Investigative Site, Oxnard, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, San Diego, California
  - Syrentis Clinical Research, 1401 N Tustin Ave, Suite 130, Santa Ana, California
  - Novartis Investigative Site, Sebastopol, California
  - Novartis Investigative Site, Sherman Oaks, California
  - Mountain Neurological Research, 350 Market Street, Suite 316, Basalt, Colorado
  - Colorado Springs Neurological, 2312 North Nevada Avenue, Suite 100, Colorado Springs, Colorado
  - Denver Neurological Clinic, 950 E Harvard Ave, Denver, Colorado
  - Yale University, One Church Street, Suite 600, New Haven, Connecticut
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Atlantis, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research, Inc., 800 NW 17th Avenue, Delray Beach, Florida
  - Infinity Clinical Research LLC, 4925 Sheridan Street, Suite 200, Hollywood, Florida
  - Alzheimer's Research and Treatment Center, 5065 State Road 7, Suite 102, Lake Worth, Florida
  - Meridien Research, 2300 Maitland center, Pkwy Ste 230, Maitland, Florida
  - Novartis Investigative Site, Melbourne, Florida
  - Novartis Investigative Site, Merritt Island, Florida
  - Novartis Investigative Site, Miami, Florida
  - New Horizon Research Center, 11880 SW 40 St., Suite 405, Miami, Florida
  - Miami-Dade Medical Research, 8955 SW 87 CT, Suite 112, Miami, Florida
  - Novartis Investigative Site, Miami Beach, Florida
  - Compass Research, LLC,100 West Gore Street, Suite 202, Orlando, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Palm Beach Gardens, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Roskamp Institute, Inc., 2040 Whitfield Avenue, Sarasota, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Hawaii Pacific Neuroscience, 2230 Liliha st 104, Honolulu, Hawaii
  - Advanced Clinical Research, 2950 E Magic View Dr, Suite 182, Meridian, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Alexian Brothers Neuroscience, 800 Biesterfield Rd, Neuroscience Institute Brock, Elk Grove Village, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Fairway, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Boston, Massachusetts
  - QUEST Research Institute, 28595 Orchard Lake Road, Suite 301, Farmington Hills, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Rochester, Minnesota
  - Hattiesburg Clinic, 415 South 28th Avenue, Hattiesburg, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, West Long Branch, New Jersey
  - Albuquerque Neuroscience, 101 Hospital Loop ne, 209 209, Albuquerque, New Mexico
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, East Syracuse, New York
  - Novartis Investigative Site, Latham, New York
  - NYU Langone Medical Center, 145 East 32nd Street, 2nd Floor, Room 226, New York, New York
  - Novartis Investigative Site, Orangeburg, New York
  - Novartis Investigative Site, Rochester, New York
  - ANI Neurology, PLLC dba Alzhe, 7809 Sardis Road, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Tulsa Clinical Research LLC, 1705 E 19th ST., STE 406/408, Tulsa, Oklahoma
  - Summit Research Network, 2701 NW Vaughn St, Suite 350, Portland, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Jenkintown, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Abington Neurological Associate Ltd., 2325 Maryland Road, Suite 100, Willow Grove, Pennsylvania
  - Rhode Island Hospital and Memory Research Institute, 1018 Waterman Ave, East Providence, Rhode Island
  - Butler Hospital, 345 Blackstone Blvd., Providence, Rhode Island
  - Roper Hospital, 316 Calhoun Street 5th Floor, Charleston, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Bennington, Vermont
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Heidelberg West, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (9):
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Kentville, Nova Scota
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Toronto Memory Program, 1 Valleybrook Drive Suite 400, Toronto, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Santiago, Chile
- China (3):
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangdong
- Finland (2):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Turku
- France (6):
  - Novartis Investigative Site, Strasbourg, Cedex
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villeurbanne
- Germany (6):
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Siegen
- Novartis Investigative Site, Kopavogur, Iceland
- Israel (5):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan
- Japan (9):
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Osaka
- Mexico (3):
  - Novartis Investigative Site, Mexico City, Mexico CP
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacán, Sinaloa
- Netherlands (2):
  - Novartis Investigative Site, 's-Hertogenbosch, North Brabant
  - Novartis Investigative Site, Amsterdam
- Portugal (4):
  - Novartis Investigative Site, Torres Vedras, Lisbon District
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
- Inspira Clinical Research, Ave Hostos 405, San Juan, Puerto Rico
- Novartis Investigative Site, Singapore, Singapore
- South Africa (3):
  - Novartis Investigative Site, Rosebank, Johannesburg
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, ZAF
- South Korea (4):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Terrassa, Barcelona
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Basel, CH
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
- Taiwan (3):
  - Novartis Investigative Site, Kaoshiung
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taipei
- United Kingdom (10):
  - Novartis Investigative Site, Exeter, Devon
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Avon
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8970 participants were screened
Period: Overall Study
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Started | 456 | 233 | 456
Patient Misrandomized | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 456 | 233 | 456
Not completed — Study terminated by Sponsor | 424 | 222 | 438
Not completed — Withdrawal by Subject | 18 | 7 | 13
Not completed — Adverse Event | 10 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Non-compliance with study treatment | 1 | 0 | 0
Not completed — Technical problems | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient was misrandomized and not included in the CNP520 50mg arm
Groups:
- Total: Total of all reporting groups
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo | Total
Number analyzed (Participants) | 455 | 233 | 456 | 1144
Age, Customized [Number; unit: participants]
  <=64 | 76 | 45 | 80 | 201
  65-69 | 181 | 82 | 162 | 425
  >70 | 198 | 106 | 214 | 518
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 148 | 288 | 720
  Male | 171 | 85 | 168 | 424
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 416 | 213 | 422 | 1051
  Black | 7 | 1 | 5 | 13
  Asian | 18 | 12 | 22 | 52
  Native American | 3 | 2 | 1 | 6
  Pacific Islander | 2 | 1 | 0 | 3
  Other | 4 | 2 | 0 | 6
  Unknown | 5 | 2 | 6 | 13
Baseline cognitive scale assessment [Mean (Standard Deviation); unit: scores on a scale] — APCC(API Preclinical Composite Cognitive Battery) is a composite score derived from RBANS(Repeatable Battery for Assessment of Neurological Status), MMSE(Mini-Mental State Examination) and the Raven's Progressive Matrices; scores: 0-100/higher scores=better cognitive performance. RBANS is a tool to detect/characterize neurocognitive dementia changes in 5 neurocognitive domains; scores: 40-160/higher scores=better cognitive functioning. Clinical Dementia Rating Sum of Boxes(CDR-SOB) measures cognition+functioning in 6 domains; scores: 0-18/higher scores indicate greater disease severity
  scores on a scale
    APCC score | 74.6 (6.68) | 75.8 (6.81) | 74.9 (7.16) | 75.0 (6.91)
    RBANS Total | 100.5 (11.96) | 102.0 (12.09) | 100.7 (12.42) | 100.9 (12.18)
    CDR-SOB | 0.19 (0.389) | 0.16 (0.358) | 0.14 (0.358) | 0.16 (0.371)

OUTCOME MEASURES:

1. Primary Outcome: Time to Event (Diagnosis of Mild Cognitive Impairment or Dementia, Due to Alzheimer's Disease (AD))
Description: Event was defined as the first confirmed diagnosis of MCI due to Alzheimer's disease (AD) or dementia due to AD (whichever occurred first) after adjudication by the progression adjudication committee (PAC) as triggered either by an investigator diagnosis or an increase in the Clinical Dementia Rating (CDR) global score. An event had to be confirmed by the PAC at two consecutive visits. In case no confirmed event was observed for a participant, the observation was censored, and the censoring date was defined as the last date where the diagnostic classification was assessed. The Study was terminated and only confirmed events collected up to the data cut-off point were counted. Due to the early termination of the study only a small number of events were observed and time-to-event could not be analyzed. Kaplan-Meyer (KM) estimates were provided to estimate probability that a subject would have an event prior to the specified visit.
Time Frame: Baseline to last cognitive assessment performed (up to day 648)
Population: Safety analysis set; n=number of participants at risk to experience an event at the time-point
Measure: Number (95% Confidence Interval); unit: probability of an event
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 455 | 233 | 456
probability of an event
  Week 26 n=232,123,250: number analyzed (Participants) | 232 | 123 | 250
  Week 26 n=232,123,250 | 0.99 [0.96 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [0.97 to 1.00]
  Week 52 n=52,24,57: number analyzed (Participants) | 52 | 24 | 57
  Week 52 n=52,24,57 | 0.97 [0.94 to 0.99] | 0.99 [0.92 to 1.00] | 0.99 [0.96 to 1.00]
  Week 78 n=6,2,2: number analyzed (Participants) | 6 | 2 | 2
  Week 78 n=6,2,2 | 0.97 [0.94 to 0.99] | 0.99 [0.92 to 1.00] | 0.97 [0.88 to 0.99]

2. Primary Outcome: Change in the Alzheimer's Prevention Initiative Composite Cognitive (APCC) Test Score
Description: APCC is a composite score derived from the specific scores from the Repeatable Battery for the Assessment of Neurological Status (RBANS), Mini-Mental State Examination (MMSE) and the Raven's Progressive Matrices. The APCC score is a weighted score with ranges from from 0 to 100 where higher scores correspond to better cognitive performance.
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: Safety analysis set - only participants with a value at both Baseline and that visit are included. Last on-treatment is the last assessment before or at last day on study drug + 31 days. Last off-treatment is the last assessment after last day on study drug + 31 days.
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 269 | 144 | 275
Total scores
  Week 26 n=160,79,162: number analyzed (Participants) | 160 | 79 | 162
  Week 26 n=160,79,162 | -3.1 (5.20) | -2.9 (5.00) | -1.7 (4.44)
  Last on-treatment n=269,144,275 | -2.2 (4.88) | -0.8 (4.67) | -1.3 (5.21)
  Last off-treatment n=255,124,260: number analyzed (Participants) | 255 | 124 | 260
  Last off-treatment n=255,124,260 | -0.8 (4.56) | -0.8 (4.38) | -0.8 (4.64)

3. Secondary Outcome: Change in Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) Score
Description: The CDR was obtained through semi-structured interviews of participants and informants, and cognitive functioning was rated on a 5-point scale of functioning in six domains: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care. The CDR global score ranged from zero to three, while the CDR-SOB was the sum of the ratings from the six domains, ranging from 0 to 18 with a minimum increment of 0.5. Higher scores indicated greater disease severity
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 265 | 144 | 267
Scores on a scale
  Week 26 n=160,78,160: number analyzed (Participants) | 160 | 78 | 160
  Week 26 n=160,78,160 | 0.17 (0.606) | 0.20 (0.451) | 0.08 (0.385)
  Last on-treatment n=265,144,267 | 0.15 (0.557) | 0.08 (0.449) | 0.10 (0.468)
  Last off-treatment n=254,117,256: number analyzed (Participants) | 254 | 117 | 256
  Last off-treatment n=254,117,256 | 0.09 (0.525) | 0.07 (0.401) | 0.10 (0.565)

4. Secondary Outcome: Change in the Total and Index Scores of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: Repeatable Battery for the Assessment of Neurological Status (RBANS) is a clinical tool designed to detect and characterize the earliest neurocognitive changes associated with dementia. The RBANS generates age-adjusted index scores for five neurocognitive domains: Immediate Memory, Visuospatial/Constructional, Language, Attention and Delayed Memory, which are used to calculate a Total Scale Index score. Index scores and total score range from 40 to 160 and a higher score indicates better cognitive functioning.
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 356 | 183 | 353
scores
  Total Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Total Week 26 n=162,81,162 | -5.8 (8.54) | -6.3 (8.58) | -3.4 (8.35)
  Total Last on-treatment n=356,183,353 | -3.4 (8.66) | -3.5 (8.87) | -0.5 (8.88)
  Total Last off-treatment n=259,125,265: number analyzed (Participants) | 259 | 125 | 265
  Total Last off-treatment n=259,125,265 | -1.3 (8.12) | -2.4 (9.55) | -1.9 (8.56)
  Immediate memory - Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Immediate memory - Week 26 n=162,81,162 | -9.8 (11.85) | -9.7 (12.10) | -5.2 (11.26)
  Immediate memory - Last on-treatment n=347,183,353: number analyzed (Participants) | 347 | 183 | 353
  Immediate memory - Last on-treatment n=347,183,353 | -5.9 (13.01) | -4.0 (13.54) | -1.1 (13.04)
  Immediate memory - Last off-treatment n=259,125,266: number analyzed (Participants) | 259 | 125 | 266
  Immediate memory - Last off-treatment n=259,125,266 | -3.1 (12.50) | -4.8 (13.52) | -3.0 (13.00)
  Visuospatial Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Visuospatial Week 26 n=162,81,162 | -5.6 (15.11) | -5.4 (15.51) | -2.6 (15.26)
  Visuospatial Last on-treatment n=347,183,353: number analyzed (Participants) | 347 | 183 | 353
  Visuospatial Last on-treatment n=347,183,353 | -3.7 (14.90) | -3.8 (15.14) | -1.2 (13.95)
  Visuospatial Last off-treatment n=259,125,266: number analyzed (Participants) | 259 | 125 | 266
  Visuospatial Last off-treatment n=259,125,266 | -1.5 (14.87) | -0.7 (14.37) | -1.2 (14.56)
  Language Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Language Week 26 n=162,81,162 | -0.8 (11.48) | -1.8 (11.05) | -3.1 (11.07)
  Language Last on-treatment n=347,183,353: number analyzed (Participants) | 347 | 183 | 353
  Language Last on-treatment n=347,183,353 | -0.3 (11.95) | -1.7 (11.69) | -1.3 (12.58)
  Language Last off-treatment n=259,125,265: number analyzed (Participants) | 259 | 125 | 265
  Language Last off-treatment n=259,125,265 | -1.0 (10.93) | -2.0 (12.68) | -3.4 (11.47)
  Attention Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Attention Week 26 n=162,81,162 | 0.1 (11.19) | -0.1 (10.37) | 0.1 (10.56)
  Attention Last on-treatment n=347,183,353: number analyzed (Participants) | 347 | 183 | 353
  Attention Last on-treatment n=347,183,353 | 0.0 (11.30) | 0.0 (10.68) | 0.7 (10.99)
  Attention Last off-treatment n=259,125,265: number analyzed (Participants) | 259 | 125 | 265
  Attention Last off-treatment n=259,125,265 | 1.6 (11.59) | 1.7 (10.65) | 1.1 (9.81)
  Delayed memory - Week 26 n=162,81,162: number analyzed (Participants) | 162 | 81 | 162
  Delayed memory - Week 26 n=162,81,162 | -5.5 (11.54) | -5.0 (11.68) | -2.1 (11.69)
  Delayed memory - Last on-treatment n=346,183,353: number analyzed (Participants) | 346 | 183 | 353
  Delayed memory - Last on-treatment n=346,183,353 | -3.0 (11.58) | -2.8 (10.56) | 0.8 (11.43)
  Delayed memory - Last off-treatment n=259,125,265: number analyzed (Participants) | 259 | 125 | 265
  Delayed memory - Last off-treatment n=259,125,265 | -1.0 (10.91) | -2.5 (10.34) | -0.5 (10.57)

5. Secondary Outcome: Change in the Everyday Cognition Scale (ECog-Subject) Total Scores
Description: Everyday Cognition Scale (ECog) measures cognitively-relevant everyday abilities comprised of 39 items covering 6 cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention. The questionnaire is a self-reported measure completed by both participant and study partner (informant). The total score for the 39 items ranges from 39 to 195, with greater scores indicating worse daily function.
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 266 | 143 | 268
Total scores
  Week 26 n=155,78,157: number analyzed (Participants) | 155 | 78 | 157
  Week 26 n=155,78,157 | 0.9 (7.90) | 0.2 (5.52) | 0.5 (6.76)
  Last on-treatment n=266,143,268 | 1.6 (8.03) | 0.4 (5.62) | 0.7 (8.25)
  Last off-treatment n=249,122,255: number analyzed (Participants) | 249 | 122 | 255
  Last off-treatment n=249,122,255 | -0.1 (6.49) | 0.0 (7.02) | 0.1 (7.47)

6. Secondary Outcome: Change in the Everyday Cognition Scale (ECog-Informant) Total Scores
Description: as for outcome 5
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 252 | 138 | 255
Total scores
  Week 26 n=153,76,153: number analyzed (Participants) | 153 | 76 | 153
  Week 26 n=153,76,153 | -0.3 (7.55) | 1.7 (7.77) | -1.2 (6.10)
  Last on-treatment n=252,138,255 | 0.5 (7.58) | 0.7 (8.49) | 0.2 (7.00)
  Last off-treatment n=223,113,239: number analyzed (Participants) | 223 | 113 | 239
  Last off-treatment n=223,113,239 | 0.5 (6.97) | 0.0 (6.74) | 1.2 (9.36)

7. Secondary Outcome: Number of Participants With Newly Occurring Safety MRI Abnormalities (ARIA-E, ARIA-H,White Matter Disease and Any Other MRI Abnormalities)
Description: Safety MRI included sequences necessary for ascertainment of possible ARIA-E (Amyloid Related Imaging Abnormality-Edema), ARIA-H (Amyloid Related Imaging Abnormality- Hemorrhage, including superficial siderosis and microhemorrhages), assessment of recent infarcts and white matter integrity examination (White matter disease worsening) and a general assessment of brain abnormalities.
Time Frame: Baseline up to study termination approximately 617 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 455 | 233 | 456
Participants
  Presence of ARIA-H | 0 | 0 | 0
  Questionable presence of ARIA-E | 1 | 0 | 2
  White matter disease worsening: 1-3 increase | 4 | 2 | 3
  White matter disease worsening: 4- - >8 increase | 0 | 0 | 0
  White matter disease worsening >8 | 0 | 0 | 0
  Any other MRI abnormalities | 1 | 0 | 1

8. Secondary Outcome: Annualized Percent Change on Volume of Brain Regions
Description: Annualized % change from baseline in volume of specific brain regions of interest (ROIs): whole brain (WB), hippocampus (Hip), and lateral ventricles (LV). Annualized percentage change was calculated as (percentage per participant / time interval (in days)) x 365.25. Time interval (in days) was derived as date of current MRI assessment on study drug - date of baseline MRI assessment + 1.
Time Frame: Baseline to Week 26, Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of volume change
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 179 | 85 | 182
Percentage of volume change
  WB Week 26 n=169,83,169: number analyzed (Participants) | 169 | 83 | 169
  WB Week 26 n=169,83,169 | -1.1016 (1.03196) | -0.9348 (0.85477) | -0.5552 (1.21385)
  WB Last on-treatment n=179,85,182 | -1.0427 (0.93751) | -0.9205 (0.75633) | -0.5378 (1.09542)
  WB Last off-treatment n=72,44,81: number analyzed (Participants) | 72 | 44 | 81
  WB Last off-treatment n=72,44,81 | -0.6984 (0.73644) | -0.9188 (0.94516) | -0.5811 (0.75412)
  Hip Week 26 n=169,83,169: number analyzed (Participants) | 169 | 83 | 169
  Hip Week 26 n=169,83,169 | -2.0993 (2.77159) | -1.9100 (2.31406) | -1.2113 (2.71764)
  Hip Last on-treatment n=179,85,182 | -2.0052 (2.65898) | -1.7909 (2.06883) | -1.1628 (2.56183)
  Hip Last off-treatment n=72,44,81: number analyzed (Participants) | 72 | 44 | 81
  Hip Last off-treatment n=72,44,81 | -1.3755 (1.90613) | -1.2522 (2.23213) | -1.1929 (1.81333)
  LV Week 26 n=169,83,169: number analyzed (Participants) | 169 | 83 | 169
  LV Week 26 n=169,83,169 | 5.4388 (5.91870) | 5.3457 (4.67788) | 3.5415 (4.75268)
  LV Last on-treatment n=179,85,182 | 5.0974 (5.31542) | 5.0822 (3.88165) | 3.4582 (4.35888)
  LV Last off-treatment n=72,44,81: number analyzed (Participants) | 72 | 44 | 81
  LV Last off-treatment n=72,44,81 | 4.0014 (4.29087) | 3.9355 (5.17657) | 3.3851 (3.38576)

9. Secondary Outcome: Change in CSF Levels of Amyloid Beta 40 (Aβ40)
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): Amyloid Beta 40 (Aβ40)
Time Frame: Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 16 | 5 | 14
ng/mL
  AB40 Last on-treatment n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  AB40 Last on-treatment n=1,0,1 | -7.320 |  | -0.760
  AB40 Last off-treatment n=16,5,13: number analyzed (Participants) | 16 | 5 | 13
  AB40 Last off-treatment n=16,5,13 | -1.492 (1.9263) | 0.804 (1.9220) | -1.172 (1.7408)

10. Secondary Outcome: Change in CSF Levels of Amyloid Beta 42 (Aβ42)
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): Amyloid Beta 42 (Aβ42).
Time Frame: Baseline to Last on-treatment (Day 547) and Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 16 | 5 | 13
pg/mL
  AB42 Last on-treatment n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  AB42 Last on-treatment n=1,0,1 | -366.200 |  | -61.300
  AB42 Last off-treatment n=16,5,13 | 20.431 (74.5595) | -68.660 (62.8505) | 21.246 (104.3395)

11. Secondary Outcome: Change in Neurofibrillary Tangle Burden as Measured by Standardized Uptake Ratio (SUVR) of PET Scans With Tau Radiotracer (Where Available)
Description: To demonstrate the effects of CNP520 vs placebo on Alzheimer's Disease-related biomarkers
Time Frame: Baseline to Months 24 and 60
Population: No available data since no post-baseline (month 24 and 60) PET scan could be obtained due to the early termination of the trial.
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change in Amyloid Deposition as Measured by Standardized Uptake Ratio (SUVR) of Positron Emission Tomography (PET) Scan With Amyloid Radiotracer
Description: To demonstrate the effects of CNP520 vs placebo on Alzheimer's Disease-related biomarkers
Time Frame: Baseline to Months 24 and 60
Population: as for outcome 11
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change in CSF Levels of Total Tau and Phosphorylated Tau
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): total tau protein and phosphorylated tau protein levels
Time Frame: Baseline to Last on-treatment (Day 547) Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 16 | 5 | 13
pg/mL
  Total tau - Last on-treatment n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  Total tau - Last on-treatment n=1,0,1 | 40.000 |  | -12.600
  Total tau - Last off-treatment n=16,5,13 | -22.119 (28.6218) | -3.320 (21.1548) | -3.238 (23.4442)
  Phosphorylated tau - Last on-treatment n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  Phosphorylated tau - Last on-treatment n=1,0,1 | -2.360 |  | -0.550
  Phosphorylated tau - Last off-treatment n=16,5,13 | -1.849 (2.3397) | -0.852 (2.7005) | 0.065 (1.3032)

14. Secondary Outcome: Change in Serum Neurofilaments
Description: Alzheimer's Disease-related biomarkers analyzed in blood serum: light chain neurofilaments (NfL)
Time Frame: Baseline to Week 26, baseline to Last on-treatment (Day 547) Baseline to Last off-treatment (Day 648)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 33 | 17 | 40
pg/mL
  Week 26 n=33,17,38: number analyzed (Participants) | 33 | 17 | 38
  Week 26 n=33,17,38 | 0.622 (4.5576) | 0.901 (4.6732) | -5.731 (40.9042)
  Last on-treatment n=33,15,40: number analyzed (Participants) | 33 | 15 | 40
  Last on-treatment n=33,15,40 | 0.932 (4.2494) | 0.041 (3.4144) | -5.771 (39.8254)
  Last off-treatment n=5,2,1: number analyzed (Participants) | 5 | 2 | 1
  Last off-treatment n=5,2,1 | -2.764 (3.0981) | 7.350 (9.5884) | 3.880

15. Secondary Outcome: Number of Suicidal Ideation or Behavior Events
Description: Prospective suicidality assessment was performed with the use of Columbia-Suicide Severity Rating Scale (C-SSRS), a questionnaire using a detailed branched logic algorithm evaluating participant's suicidality ideation and behavior. Answer "yes" on item 4 or 5 of the Suicidal Ideation section or "yes" on any item of the Suicidal Behavior section was considered positive.
Time Frame: Baseline up to study termination approximately 617 days
Population: Safety analysis set which includes only participants with events
Measure: Number; unit: events
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
Number analyzed (Participants) | 455 | 233 | 456
events
  Any suicidal ideation n=13,3,9: number analyzed (Participants) | 13 | 3 | 9
  Any suicidal ideation n=13,3,9 | 25 | 6 | 12
  Any suicidal behavior n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  Any suicidal behavior n=1,0,1 | 1 |  | 1

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 31 days of washout period for a maximum duration of 617 days.
Arm/Group | CNP520 50 mg | CNP520 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/455 | 0/233 | 0/456
Serious Adverse Events (participants affected / at risk) | 15/455 | 9/233 | 15/456
Other Adverse Events (participants affected / at risk) | 137/455 | 62/233 | 89/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNP520 50 mg (N=455) | CNP520 15 mg (N=233) | Placebo (N=456)
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CNP520 50 mg (N=455) | CNP520 15 mg (N=233) | Placebo (N=456)
Bronchitis (Infections and infestations) | 6 | 7 | 4
Nasopharyngitis (Infections and infestations) | 22 | 9 | 11
Upper respiratory tract infection (Infections and infestations) | 18 | 5 | 16
Urinary tract infection (Infections and infestations) | 8 | 8 | 7
Fall (Injury, poisoning and procedural complications) | 11 | 7 | 5
Weight decreased (Investigations) | 19 | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 2 | 4
Dizziness (Nervous system disorders) | 14 | 7 | 8
Headache (Nervous system disorders) | 12 | 8 | 15
Abnormal dreams (Psychiatric disorders) | 18 | 7 | 3
Anxiety (Psychiatric disorders) | 21 | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 12 | 16

LIMITATIONS AND CAVEATS:
The study was terminated due to safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03131453/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03131453/SAP_001.pdf